CLINICAL TRIAL: NCT03825562
Title: Acceptance and Value Based Based Methods in Increasing Wellbeing of Adolescents With Type 1 Diabetes / Hyväksyntä- ja Arvopohjaiset menetelmät Diabetesta Sairastavien Nuorten Hyvinvoinnin edistämisessä
Brief Title: Acceptance and Value Based Methods in Increasing Wellbeing of Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Finland Hospital District (Other)
Collaborators: University of Jyvaskyla (Other); Finnish Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dnro 7U/2015
Record Dates: First submitted 2017-01-30; First posted 2019-01-31 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2019-05

CONDITIONS: Diabetes
Keywords: type 1 diabetes; ACT; adolescents; value based methods; acceptance
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- research group (Experimental): Research group is attending the ACT intervention first and from before and afte measurement are compared to the control group
  Interventions: Behavioral: acceptance and commitment therapy, ACT
- control group (Active Comparator): Control group is offered to attend the intervention afterwards
  Interventions: Behavioral: acceptance and commitment therapy, ACT

INTERVENTIONS:
Behavioral: acceptance and commitment therapy, ACT

SUMMARY:
The aim of the study is to study how using acceptance and value based group intervention helps the wellbeing of teenagers with type in diabetes.

The investigators created an ACT-group intervention consisting of five sessions, based on earlier research. 12-16 years- old diabetics who are treated at KSSHP pediatric policlinic are invited to join the groups. The participants are randomized to research and control groups. The HbA1c-level is monitored for both groups as well as the psychological flexibility, diabetes related acceptance, depression and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes

Exclusion Criteria:

* weekly psychiatric appointments

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-10; Primary Completion 2020-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Glycemic control | up to 8 months
  HbA1c

SECONDARY OUTCOMES:
Quality of life assessed by KINDL-r Questionnaire | up to 8 months
  To measure the quality of life the Revised Children's Quality of Life Questionnaire is used. The KINDLr is a generic instrument for assessing Health-Related Quality of Life in children and adolescents aged 3-17 years (Ravens-Sieberer & Bullinger, 1998). In this study, we use the generic, youth-specific, mode of the questionnaire consisting of 24 questions and the diabetes specific module consisting of 17 questions. The answers are given on the Likers Scale from 1-5. The generic mode consists of 6 sub-scales: physical well-being, emotional well-being, self-esteem, social contacts and school. The six sub-scales are combined to form a total score of maximum 120. The maximum score in diabetes specific module is 85. Higher scores indicate better quality of life.
Diabetes Related Psychological flexibility assessed by DAAS | up to 8 months
  To measure diabetes related acceptance skills the DAAS-questionnaire (The Diabetes Acceptance and Action Scale for Children and Adolescents) is used. A questionnaire is developed to measure the diabetes related psychological flexibility (Greco & Hart, 2005). Questionnaire consists of 42 questions and responses are given on Likert scale from 0-4. The maximum score in the questionnaire is 168. The higher sum in the questionnaire refers to higher psychological flexibility, better acceptance of diabetes and action.
Depressive symptoms assessed by RBDI | up to 8 months
  To measure the depressive symptoms and anxiety the RBDI-questionnaire (Revised Beck Depression Inventory) is used. RBDI is a Finnish version of The Beck Depression Inventory (Beck & Beck, 1972). It consists of 13 questions measuring depressive symptoms and one question measuring anxiety. In each question there are five possible answers to choose and scores are given from 0 to 3. The maximum score for measuring depressive symptoms is 39 and the maximum score for the question measuring anxiety is 3. Higher scores means more symptoms of depression or anxiety.
Psychological flexibility assessed by CAMM | up to 8 months
  To asses psychological flexibility CAMM (The Child and Adolescent Mindfulness measure) is used. CAMM-questionnaire was developed to measure the mindfulness and acceptance skills and it assesses the degree to which children and adolescents observe internal experiences, act with awareness, and accept internal experiences without judging them (Greco, Baer, & Smith, 2011). The 10-question version is used. The answers are given on Likert scale 0-4, from never true to always true. Maximum score is 40. Higher scores indicate higher levels of mindfulness and acceptance.

CONTACTS AND LOCATIONS:
Overall Officials: Raimo Lappalainen, PhD, Study Director — supervisor
Locations (1):
- Iina Alho, Jyväskylä, Finland

IPD SHARING:
Plan to Share IPD: No